CLINICAL TRIAL: NCT03295565
Title: A Randomized, Open Label, Phase IIB Trial of Optimal Sequencing of Treatment Options for Poor Risk Metastasized Castration Resistant Prostate Cancer Previously Treated With Docetaxel
Brief Title: Optimal Sequencing of Treatment Options for Poor Risk mCRPC Previously Treated With Docetaxel
Acronym: OSTRICh
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: m16OST
Record Dates: First submitted 2017-07-17; First posted 2017-09-28 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer Metastatic; Metastasis
Keywords: Sequencing; cabazitaxel; abiraterone; enzalutamide; clinical benefit rate; docetaxel; second line treatment
MeSH Terms: conditions — Neoplasm Metastasis | interventions — cabazitaxel; abiraterone; enzalutamide

STUDY DESIGN:
Intervention Model Description: randomized, open label, Phase IIB trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Cabazitaxel (Active Comparator): Cabazitaxel 25mg/m2 IV, once every 3 weeks
  Interventions: Drug: Cabazitaxel
- B: Abiraterone OR Enzalutamide (Active Comparator): At physician's discretion:
  Abiraterone 1000mg oral, taken daily Prednisone 5mg oral, 2 times a day OR Enzalutamide 160mg oral taken daily
  Interventions: Drug: Abiraterone; Drug: Enzalutamide

INTERVENTIONS:
Drug: Cabazitaxel — Cabazitaxel 25mg/m2 IV, once every 3 weeks
  Other Names: No other intervention names
  Arms: A: Cabazitaxel
Drug: Abiraterone — Abiraterone 1000mg oral, taken daily + Prednisone 5mg oral, 2 times a day
  Other Names: No other intervention names
  Arms: B: Abiraterone OR Enzalutamide
Drug: Enzalutamide — Enzalutamide 160mg oral taken daily
  Other Names: No other intervention names
  Arms: B: Abiraterone OR Enzalutamide

SUMMARY:
Rationale:

The aim of this study is to identify the optimal second line treatment option for patients with a poor prognosis metastasized Castration Resistant Prostate Cancer (mCRPC) with respect to Clinical Benefit Rate (CBR) rate and quality of life.

Objective:

The primary endpoint is CBR in mCRPC patients with poor prognostic features and previously treated with docetaxel, randomized between cabazitaxel (Arm A) and novel hormonal agents (abiraterone OR enzalutamide) as second-line therapy (Arm B).

Intervention:

Patients in Arm A will receive cabazitaxel and prednisone and patients in Arm B will receive abiraterone and prednisone OR enzalutamide.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Treatment regimens evaluated in this trial are used in common mCRPC treatment practice and are reimbursed. Risk of side effects or death as a result of treatment is not affected by the trial design. At baseline, prior to each treatment cycle and at end of treatment, patients are requested to visit the out-patient clinic, where a physical exam will be performed in combination with vena puncture for blood analysis. Radiological evaluation will be performed at base line, after 3 months of treatment and at end of treatment. All above mentioned interventions can be considered as standard practice. Patients are requested to fill out QoL and pain/analgesic use questionnaires at base line, prior to each cycle and at end of treatment.

DETAILED DESCRIPTION:
Rationale:

The aim of this study is to identify the optimal second line treatment option for patients with a poor prognosis metastasized Castration Resistant Prostate Cancer (mCRPC) with respect to Clinical Benefit Rate (CBR) rate and quality of life.

Objective:

The primary endpoint is CBR in mCRPC patients with poor prognostic features and previously treated with docetaxel, randomized between cabazitaxel (Arm A) and novel hormonal agents (abiraterone OR enzalutamide) as second-line therapy (Arm B).

Study design:

a prospective, multicenter, national, randomized, open label phase IIB study. Study population: Males over 18 years with mCRPC, previously treated with docetaxel and features of poor prognostic disease; including duration of response to androgen deprivation shorter than one year, liver metastases, disease progression during docetaxel treatment or within 6 months after docetaxel treatment completion.

Intervention:

Patients in Arm A will receive cabazitaxel and prednisone and patients in Arm B will receive abiraterone and prednisone OR enzalutamide.

Main study parameters/endpoints: Primary endpoint: Clinical benefit rate (CBR). Secondary endpoints include: formal comparison of the CBR in both study arms, Time To Symptomatic Progression (TTSP), Time To PSA (prostate specific antigen), Progression (TTPP), and Time To Radiologic Progression (TTRP), progression free survival, overall survival, safety/ toxicity profile and Quality of Life (QoL) and pain response.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Treatment regimens evaluated in this trial are used in common mCRPC treatment practice and are reimbursed. Risk of side effects or death as a result of treatment is not affected by the trial design. At baseline, prior to each treatment cycle and at end of treatment, patients are requested to visit the out-patient clinic, where a physical exam will be performed in combination with vena puncture for blood analysis. Radiological evaluation will be performed at base line, after 3 months of treatment and at end of treatment. All above mentioned interventions can be considered as standard practice. Patients are requested to fill out QoL and pain/analgesic use questionnaires at base line, prior to each cycle and at end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of prostate adenocarcinoma.
2. Able and willing to provide informed consent and to comply with the study procedures
3. Age ≥18
4. Evidence of bone, visceral and/or lymph node metastases on bone scan, CT-scan or MRI.
5. Must have received at least one prior regimen of docetaxel treatment for at least 12 weeks (four courses) and no other prostate cancer treatments between docetaxel and randomization, other than prednisone.
6. Continued androgen deprivation therapy either by luteinizing hormone release hormone (LHRH) agonist/ antagonist or orchiectomy.
7. Treatment with curative intent is not an option and patient has an indication for systemic treatment as judged by the medical care provider
8. Evidence of progressive metastatic disease by PSA progression (Prostate Cancer Working Group 3 (PCWG3) criteria20: at least 2 rises at a minimum of 1-week intervals. The first PSA value must be ≥ 2 ng/ml) and/or radiological progression as evaluated by chest, abdominal, or pelvic CT/MRI scan and/or bone scan within 28 days of registration (see Appendix III)
9. Poor prognosis disease as defined by any of the following:

   1. The presence of liver metastases AND/OR
   2. Development of castration-resistance within 12 months of orchiectomy or commencement of LHRH antagonist/agonist for metastatic disease AND/OR
   3. Progressive disease during docetaxel treatment or <6 months after completion of docetaxel treatment
10. World Health Organization Performance Status (WHO PS) 0-2.
11. Serum testosterone < 50 ng/dL (< 1.7 nmol/L) within 28 days before treatment group allocation
12. At least 21 days have passed since completing radiotherapy (exception for a single fraction of ≤ 800 centi-Gray (cGy) to a restricted field or limited-field radiotherapy to non-marrow bearing area such as an extremity or orbit: at least 7 days prior to randomization).
13. At least 21 days have passed since major surgery.
14. Neuropathy ≤ grade 1 at the time of registration.
15. Has recovered from all therapy-related toxicity to ≤ grade 2 (except alopecia, anemia and any signs or symptoms of androgen deprivation therapy) at the time of registration.
16. Eligible for cabazitaxel, abiraterone acetate or enzalutamide as per standard of care practices.
17. Men treated with cabazitaxel should use effective contraception throughout treatment and are recommended to continue this for up to 6 months after the last dose of cabazitaxel. Due to potential exposure via seminal liquid, men treated with cabazitaxel should prevent contact with the ejaculate by another person throughout treatment. Men being treated with cabazitaxel are advised to seek advice on conservation of sperm prior to treatment.

Exclusion Criteria:

1. Histologic evidence of small cell/neuroendocrine prostate cancer
2. Any treatment other than prednisone between docetaxel and cabazitaxel/abiraterone OR enzalutamide sequence
3. Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus).
4. History of severe hypersensitivity reaction (≥ grade 3) to docetaxel, abiraterone or enzalutamide (whichever applies).
5. History of severe hypersensitivity reaction (≥ grade 3) to polysorbate 80 containing drugs.
6. Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who are already on these treatments).
7. Patients who have a concurrent yellow fever vaccination (several weeks before start of treatment) must be excluded.
8. Dementia, altered mental status, or any psychiatric condition, if this is in conflict with the study.
9. Unable to swallow a whole tablet or capsule
10. Contraindications to the use of corticosteroid treatment
11. Symptomatic peripheral neuropathy Grade ≥2 (see Appendix VIII).
12. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured and needing no subsequent therapy.
13. Inadequate organ and bone marrow function as evidenced by:

    1. Hemoglobin <10.0 g/dL
    2. Absolute neutrophil count <1.5 x 109/L
    3. Platelet count < 100 x 109/L
    4. aspartate aminotransferase (AST)/ serum glutamate oxaloacetate transaminase (SGOT) and/ or Alanine Aminotransferase (ALT)/ serum glutamate pyruvate transaminase (SGPT) > 1.5 x (upper limit of normal) ULN Total bilirubin >1 x ULN (except for patients with documented Gilbert's disease).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Clinical benefit rate | From start treatment until 12 weeks of treatment
  • To assess the Clinical Benefit Rate (CBR) in patients with mCRPC and poor prognostic factors treated with cabazitaxel (Arm A) or novel hormonal agents (abiraterone OR enzalutamide) as second-line therapy (Arm B) who have been treated with docetaxel.

SECONDARY OUTCOMES:
Comparing clinical benefit rate in arm A and arm B | From start treatment until 12 weeks of treatment
  • To formally compare the Clinical Benefit Rate (CBR) in both study arms A and B.
Duration of treatment | for each patient; until end of treatment (for Arm A max 30 weeks, for Arm B max 24 months)
  • To determine duration of treatment (DOT) in mCRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy and for those who cross over to the other study arm as a third-line therapy.
Progression free survival | for each patient; until progression or through study completion (max 24 months)
  • To determine the Progression Free Survival (PFS) of mCRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy and for those who cross over to the other study arm as a third-line therapy.
Overall survival | for each patient; until death or end of trial (max 24 months)
  • To determine the Overall Survival (OS) of mCRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy.
(serious) adverse events according to the ctcae v4.03: number of incidents, number of participants with (S)AE's | for each patient: until 28 days after the last treatment
  • To evaluate safety and toxicity profile of cabazitaxel and novel hormone agents (abiraterone OR enzalutamide) as a second line treatment.
Quality of Life assesed by the FACT-P questionnaire | for each patient; until start of the next therapy, death or end of trial (max 24 months)
  • Quality of Life (QoL) as assessed by Fundamental Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire in metastatic CRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy.
Quality of Life as assessed by the BPI-S questionnaire | for each patient; until start of the next therapy, death or end of trial (max 24 months)
  • Quality of Life (QoL) as assessed Brief Pain Inventory-Short form (BPI-S) questionnaire in metastatic CRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy.
Use of pain medication, assessed by a questionnaire about opiate use. | for each patient; until start of the next therapy, death or end of trial (max 24 months)
  Use of pain medication, assessed by a questionnaire about opiate use in metastatic CRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy.
Time to symptomatic progression | for each patient: until symptomatic progression or through study completion (max 24 months)
  Time To Symptomatic Progression (TTSP) in CRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy and for those who cross over to the other study arm as a third-line therapy.
Time to PSA progression | for each patient: until PSA progression or through study completion (max 24 months)
  Time To PSA Progression (TTPP) in mCRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy and for those who cross over to the other study arm as a third-line therapy.
Time to Radiological progression | for each patient: until radiological progression or through study completion (max 24 months)
  Time To Radiological Progression (TTRP) in mCRPC patients treated with cabazitaxel or novel hormone agents (abiraterone OR enzalutamide) as second-line therapy and for those who cross over to the other study arm as a third-line therapy.
PSA>50% decrease | for each patient; from baseline until end of trial (max 24 months)
  Rate of PSA>50% decrease from baseline

OTHER OUTCOMES:
Exploratory objectives; neutrophil to lymphocyte ratio | For each patient: until the end of treatment, Arm A max 30 weeks, Arm B max 24 months
  Prostate cancer is a very diverse disease and there is a need for more personalized treatment than offered nowadays. Therefore, three biomarker studies are included in this randomized trial. The value of the neutrophil to lymphocyte ratio will be measured in all patients, to try to find a predictive value
Exploratory objectives; number of mutations in 73 genes from cell-free DNA | For each patient: until the end of treatment, Arm A max 30 weeks, Arm B max 24 months
  We will draw blood from patients to measure mutations in 73 prostate cancer-related genes out of cell-free DNA. The goal again is to find a predictive value in these DNA mutations and to be able to give more personalized treatment.
Exploratory objectives; epigenetics-based biomarker discovery using cfDNA | For each patient: until end of treatment (max 24 months)
  We will isolate chromatinized cfDNA from serum samples of all patients in this trial. Immunoprecipitation will be performed for H3K27ac after which isolated DNA fragments are sequenced, effectively sequencing the enriched functional enhancers that are detected in the serum-derived cfDNA. The aim is to identify distinct functional enhancers that enable outcome prediction.

CONTACTS AND LOCATIONS:
Locations (19):
- Netherlands (19):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Bovenij ziekenhuis, Amsterdam
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooi Ziekenhuizen, Blaricum
  - Deventer Ziekenhuis, Deventer
  - Slngeland Ziekenhuis, Doetinchem
  - Ziekenhuisgroep Twente, Hengelo
  - Spaarne Ziekenhuis, Hoofddorp
  - Dijklander ziekenhuis, Hoorn
  - Medisch Centrum leeuwarden, Leeuwarden
  - Academisch medisch centrum Maastricht, Maastricht
  - Sint Antonius ziekenhuis, Nieuwegein
  - Franciscus Gasthuis-Vlietland, Rotterdam
  - Zorgsaam Ziekenhuis, Terneuzen
  - Haga Ziekenhuis, The Hague
  - Diakonessenhuis, Utrecht
  - Universitair medisch centrum Utrecht, Utrecht
  - Viecuri medisch centrum Noord-Limburg, Venlo
  - Isala Klinieken, Zwolle